CLINICAL TRIAL: NCT06369012
Title: Randomized Trial of Mefenamic Acid Versus Tranexamic Acid in Management of Abnormal Uterine Bleeding
Brief Title: Management of Abnormal Uterine Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Rania Gamal
Record Dates: First submitted 2024-04-09; First posted 2024-04-16 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2024-04

CONDITIONS: Abnormal Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia | interventions — Mefenamic Acid; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A : Mefenamic acid (Active Comparator): About 65 women will take Mefenamic acid tablets orally, 3 timed per day.This regiment can be repeated for at least three attacks of Abnormal Uterine Bleeding.
  (Mefenamic acid manufactured by JPI pharmaceutical company)
  Interventions: Drug: Mefenamic acid 500 mg
- Group B: Tranexamic acid (Active Comparator): About 65 women will take Tranexamic acid capsules orally, 3 time per day .This regiment can be repeated for at least three attacks of Abnormal Uterine Bleeding.
  (Tranexamic acid manufactured by AMOUN pharmaceutical company)
  Interventions: Drug: Mefenamic acid 500 mg

INTERVENTIONS:
Drug: Mefenamic acid 500 mg — To compare the effectiveness of mefenamic acid versus tranexamic acid in the management of abnormal uterine bleeding.
  Other Names: Tranexamic Acid 500 mg

SUMMARY:
Abnormal uterine bleeding "AUB" describes all abnormal forms of menstrual bleeding which may result from several causes including anovulation, problems related to pregnancy, infections, vaginal and cervical abnormalities, uterine pathologies including benign and malignant tumors, coagulopathies, endocrine disorders, trauma, foreign bodies, systemic diseases and iatrogenic causes. AUB may be clinically presented by menorrhagia, metrorrhagia or menometrorrhagia. It's the most common complaint for the reproductive age females and accounts for 33% of female patients referred to gynecologists

DETAILED DESCRIPTION:
Menorrhagia, if repeated, causes a decrease in iron reserve and anemia and subsequently, anemia causes psychological and cardiac complications and dysfunction in other organs. So, paying attention to menorrhagia and its treatment can lead to lower morbidity in reproductive aged women. It is worth noticing that most of the iron deficient anemia morbidities are the result of more than 60 ml bleeding per cycle.

The evaluation of the actual bleeding volume is not an easy task because women's evaluation of their own bleeding volume is not reliable. 25% of the women who consider their bleeding level as high had menstrual bleeding less than 35 ml. The estimation of blood loss volume was done based on the number of pads or tampons soaking per day or per cycle. The patient's estimations of the bleeding volumes are not accurate and reliable because they are not well aware of the normal range of bleeding and their evaluations are inexact.

Ideally, a noninvasive investigation is preferred to an invasive one and also an economical investigation preferred to an expensive one; this applies equally to affluent countries and third world, that is why ultrasonography by any modality if available is considered to be a noninvasive procedure to investigate uterine lesions rather than hysteroscopy as a preliminary step .

Various imaging techniques are used to enable the precise localization and characterization of uterine pathology. Currently, the main diagnostic tools for AUB include ultrasonography and diagnostic hysteroscopy.

Menorrhagia is defined as complaint of heavy menstrual bleeding over several consecutive cycles. The upper limit of monthly bleeding is 80 ml per cycle, which is 2 standard deviations from the mean (mean menstrual bleeding per cycle is 36 - 52ml).

Worldwide use of hormonal therapy is based on the wrong assumption that menorrhagia happens because of imbalance in hormones and an ovulatory cycle, but the fact is most of the women with abnormal bleeding show no evidence of hormonal imbalance and based on some studies 95% have regular ovulatory cycles.

Antifibrinolytic medications, such tranexamic acid, function by inhibiting the breakdown of fibrin and are useful in the management of individuals with persistent AUB. It has been demonstrated that they can cut bleeding in these patients by 30 to 55%. For the treatment of acute AUB, experts advise utilizing tranexamic acid intravenously (IV) or orally.

In another study, the treatment of menorrhagia, by both mefenamic acid and tranexamic acid.they were beneficial in controlling menstrual blood loss with significant decrease in dysmenorrhea Minor side effects like epigastric pain, nausea, vomiting was more frequent in mefenamic acid group. Acceptability rate was high in both groups

ELIGIBILITY:
Inclusion Criteria:

* Any female patient in Child bearing period aging from 15-45 years complaining of Abnormal uterine.
* Abnormal uterine bleeding due to endometrial, uterine cavity lesions as diagnosed by TVS or bleeding tendency e.g. Thrombocytopenia, Platelets dysfunction and coagulation defects

Exclusion Criteria:

* Personal history of renal or hepatic impairment; previous thromboembolic disease, peptic ulcer.
* Females with evident drugs intake that cause AUB e.g warfarin, low molecular weight heparin.
* Vaginal, vulvar, and cervical causes of bleeding.
* Bleeding on top of Use of hormonal and non-hormonal contraception.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Bleeding Control | 1 week
  The paricipants of the study whom having abnormal uterine bleeding will be asked to take the drugs of the study to see the amount of blood will decrease or not

CONTACTS AND LOCATIONS:
Overall Officials: Omnia Bakar Bakar, Lecturer, Principal Investigator — Obstetrics and Gynecology, Faculty of Medicine, Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided